CLINICAL TRIAL: NCT01821092
Title: Horizontal and Vertical Dimensional Changes of Peri-implant Facial Bone Following Placement of T3 Implants: a 1-year Cone Beam Computed Tomography Study
Brief Title: Dimensional Changes of Peri-implant Facial Bone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Proed, Torino, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03.2013.Don Bosco.PROED
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Jaw, Edentulous, Partially
Keywords: osseointegrated Implant, bone level
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Bone-Anchored Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard implant, switching platform (Active Comparator): osseointegrated implant insertion and abutment connection Implants inserted in healed ridge, prosthetic connection with switching platform
  Interventions: Procedure: implant insertion and abutment connection; Device: osseointegrated implant
- immediate implant, switching platform (Active Comparator): osseointegrated implant insertion and abutment connection Implants inserted in immediate post-extraction sites, prosthetic connection with switching platform
  Interventions: Procedure: implant insertion and abutment connection; Device: osseointegrated implant

INTERVENTIONS:
Procedure: implant insertion and abutment connection — After implant insertion, immediate or in healed ridge, the titanium abutment with switching platform will be connected
Device: osseointegrated implant — Osseointegrated Implant Insertion
  Other Names: T3 implant, Biomet 3i

SUMMARY:
40 consecutive adult patients, requiring the insertion of dental implants in the aesthetic area (from second premolar to second premolar) will be enrolled in the study. At the time of surgery, a full thickness flap will be elevated, the implant bed will be prepared according to the manufacturer's instruction and the implants will be then seated into the bone. T0 corresponds to the time of implant insertion, T1 to the time of healing abutment's connection (T0=T1 for single stage implants), and T2 corresponds to 1-year follow-up from healing abutment's connection.

Cone Beam Computed Tomography (CBCT) scans will be taken immediately after abutment connection (T1) and 1-year after (T2). The midsagittal cut of each implant will be identified, and measurements will be made at predetermined levels. Horizontal facial bone thickness (HFBT) and Vertical facial bone level (VFBL) will be measured. HFBT will be measured at 0, 3, 6 and 9 mm apical to the implant platform. VFBL wil be the perpendicular distance from the implant platform to the most coronal point of the facial bone. Changes between T1 and T2 will be calculated.

DETAILED DESCRIPTION:
The long term results and benefit of implant insertion in the aesthetic area have been well documented.

In the past few years, facial dimensional changes to the alveolar process following implant placement are object os study for both humans and animals investigations Recent studies suggest that platform switching decreases bone loss by 30% to 50%. It seems that the creation of a biologic width affects peri-implant bone loss to a significant extent and that platform switching is effective when the mucosal thickness allows the establishment of an horizontal biologic width.

A new implant with an hybrid surface (T3) has been recently launched by Biomet 3i.Aim of the present study will be to evaluate the degree of 3D marginal bone remodelling around T3 Prevail implants.

MATERIALS & METHODS:

40 consecutive adult patients, requiring the insertion of dental implants in the aesthetic area (from second premolar to second premolar) will be enrolled in the study. At the time of surgery, a full thickness flap will be elevated, the implant bed will be prepared according to the manufacturer's instruction and the implants will be then seated into the bone. Implants can be placed both with a single-stage or two-stage procedure. Implants inserted with a two-stage procedure will be re-opened after a submerged period of three months.

T0 corresponds to the time of implant insertion, T1 to the time of healing abutment's connection (T0=T1 for single stage implants), and T2 corresponds to 1-year follow-up from healing abutment's connection.

It is supposed that the creation of the biological width starts with the healing abutment's connection.

CBCT scans will be taken immediately after abutment connection (T1) and 1-year after (T2). The midsagittal cut of each implant will be identified, and measurements will be made at predetermined levels. Horizontal facial bone thickness (HFBT) and Vertical facial bone level (VFBL) will be measured. HFBT will be measured at 0, 3, 6 and 9 mm apical to the implant platform. VFBL wil be the perpendicular distance from the implant platform to the most coronal point of the facial bone. Changes between T1 and T2 will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult patients requiring implant insertion -

Exclusion Criteria:

Pregnancy history of malignancy history of radiotherapy or chemotherapy in the last 5 years long term steroidal or antibiotic therapy

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
horizontal buccal bone thickness | 12 months after abutment connection
  On Cone Beam images, the horizontal dimensional changes of peri-implant facial bone will be measured

SECONDARY OUTCOMES:
vertical bone level | 1 year after abutment connection
  On Cone Beam images, the vertical dimensional changes of peri-implant facial bone will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Cardaropoli, DDS, Study Director — Proed, Torino, Italy
Locations (1):
- PROED, Institute for Professional Education in Dentistry, Torino, Italy

IPD SHARING:
Plan to Share IPD: No